CLINICAL TRIAL: NCT06398834
Title: Effect of Esketamine Combined With Butorphanol on Pain Management Following Video-assisted Lobectomy
Brief Title: Esketamine and Butorphanol for Post-Lobectomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second People's Hospital of Hefei City (Other)
Collaborators: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wang Hongjian, Attending doctor, Second People's Hospital of Hefei City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-keyan-007
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Esketamine; Pain; Post-thoracotomy Pain Syndrome; Thoracic Diseases
MeSH Terms: conditions — Pain; Thoracic Diseases | interventions — Esketamine; Ketamine; Butorphanol

STUDY DESIGN:
Intervention Model Description: The enrolled participants were randomly allocated to either the butorphanol group (Group B) or the esketamine combined with butorphanol group (Group BK) at a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BK (Experimental): Group BK received esketamine infusion at a rate of 0.3 mg/kg/h during surgery. Patients were provided with patient-controlled intravenous analgesia (PCIA) containing esketamine (1.5 mg/kg), butorphanol (0.15 mg/kg), and azasetron (20 mg) in a total volume of 100 ml within 48 hours after surgery.
  Interventions: Drug: Esketamine; Drug: Butorphanol
- Group B (Placebo Comparator): Group B received an equivalent volume of saline during surgery. Patients were provided with patient-controlled intravenous analgesia (PCIA) containing butorphanol (0.15 mg/kg), and azasetron (20 mg) in a total volume of 100 ml within 48 hours after surgery.
  Interventions: Drug: Butorphanol

INTERVENTIONS:
Drug: Esketamine — In the esketamine combined with butorphanol group (Group BK), patients received an intraoperative intravenous infusion of esketamine (0.3 mg/kg/h) followed by postoperative patient-controlled intravenous analgesia (PCIA) (esketamine 1.5 mg/kg + butorphanol 0.15 mg/kg + azasetron 20 mg).
  Other Names: S-Ketamine, (S)-2-(o-chlorophenyl)-2-(methylamino)cyclohexanone, L-Ketamine, (-)-Ketamine
  Arms: Group BK
Drug: Butorphanol — In the butorphanol group (Group B), patients received an equivalent volume of normal saline intraoperatively and postoperatively received PCIA without esketamine.
  Other Names: Butorphanol Tartrate, Moradol, Stadol, Torbugesic, Apo-Butorphanol, Dolorex

SUMMARY:
Post-thoracotomy pain syndrome (PTPS) affects respiratory function, hindering sputum clearance and ventilation, and represents a significant complication of thoracic surgery. The analgesic effect of esketamine combined with butorphanol in PTPS is still unclear, so this study focused on this aspect.

DETAILED DESCRIPTION:
Post-thoracotomy pain syndrome affects respiratory function, hindering sputum clearance and ventilation, and represents a significant complication of thoracic surgery. Esketamine, the left-handed optical isomer of racemic ketamine, acts as an antagonist of the N-methyl-D-aspartate (NMDA) receptor, reversing central sensitization and improving postoperative pain. Butorphanol, an opioid receptor agonist-antagonist, can alleviate visceral pain, reduce the risk of respiratory depression, and decrease postoperative morphine consumption. However, research on the analgesic effects of esketamine combined with butorphanol in thoracoscopic surgery remains limited. Therefore, this study investigated the impact of esketamine combined with butorphanol on acute pain, chronic pain, and related side effects during the perioperative period in patients undergoing video-assisted lobectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-70 years
* Classified as American Society of Anesthesiologists I-III
* Undergoing video-assisted lobectomy

Exclusion Criteria:

* Operative duration < 1 hour
* Significant comorbidities affecting vital organs such as liver, kidney, and heart
* Severe infections
* Immunodeficiency
* Coagulation disorders
* History of analgesic drug abuse
* Severe dementia or communication barriers
* Mental illnesses.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic pain | 3 months post-surgery
  To assess the patient's subjective pain intensity through the Visual Analog Pain Scale at 3 months after surgery.
  The Visual Analog Pain Scale consists of a line usually 100 mm in length. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (no pain) to the right (worst pain). The patient makes a mark reflecting his or her perception, and the distance from the left endpoint to the mark is measured, in mm.

SECONDARY OUTCOMES:
Acute pain after surgery | Within 7 days after surgery
  To assess the postoperative pain intensity of each participant through the Visual Analog Pain Scale at 6, 12 hours, and 1, 2, 3, 5, and 7 days following surgery.
  The Visual Analog Pain Scale consists of a line usually 100 mm in length. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (no pain) to the right (worst pain). The patient makes a mark reflecting his or her perception, and the distance from the left endpoint to the mark is measured, in mm.
Postoperative recovery quality | Preoperative and within 3 days after surgery
  The quality of recovery was assessed by 15-item quality of recovery (QoR-15) before surgery, on postoperative day (POD) 1, and POD 3.
  The QoR-15 is a recently developed and validated short-form postoperative QoR score. Fifteen questions assess five domains of patient-reported health status: pain, physical comfort, physical independence, psychological support and emotional state. The 11-point numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).
Intraoperative mean arterial pressure | During operation
  The patient's intraoperative mean arterial pressure was recorded to assess the effect of esketamine on the patient's vital signs.
Heart rate | During operation
  The patient's intraoperative heart rate was recorded to assess the effect of esketamine on the patient's vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Xianwen Hu, PhD, Study Chair — The Second Hospital of Anhui Medical University; Wensheng He, MD, Study Director — The Second People's Hospital of Hefei; Xin Wang, MD, Principal Investigator — The Second People's Hospital of Hefei; Zicheng Wang, MD, Principal Investigator — The Second People's Hospital of Hefei; Junbao Zhang, MD, Principal Investigator — The Second People's Hospital of Hefei
Locations (1):
- The Second People's Hospital of Hefei, Hefei, Anhui, China

REFERENCES:
- [Derived] Wang H, Wang Z, Zhang J, Wang X, Fan B, He W, Hu X. Perioperative esketamine combined with butorphanol versus butorphanol alone for pain management following video-assisted lobectomy: a randomized controlled trial. Int J Clin Pharm. 2025 Apr;47(2):452-461. doi: 10.1007/s11096-024-01850-7. Epub 2025 Jan 3. PMID 39751970